CLINICAL TRIAL: NCT03833583
Title: Transcranial Direct Current Stimulation (tDCS) to Reduce Craving in Cocaine Addiction
Brief Title: TDCS for Cocaine Addiction Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soterix Medical (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: SMIN2712-P1; HS# 18-01324, GCO# 18-1920 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2019-01-18; First posted 2019-02-07 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2019-02

CONDITIONS: Cocaine Use Disorder; Cocaine Dependence
Keywords: Transcranial Direct Current Stimulation; tDCS; Brain Stimulation; Cocaine Addiction; Drug Craving
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active tDCS (Experimental): Active Transcranial Direct Current Stimulation (tDCS), Soterix Medical mini-CT tDCS stimulator
  Interventions: Device: Soterix Medical mini-CT tDCS stimulator
- Sham tDCS (Sham Comparator): Sham (Placebo) Transcranial Direct Current Stimulation (tDCS), Soterix Medical mini-CT tDCS stimulator
  Interventions: Device: Soterix Medical mini-CT tDCS stimulator

INTERVENTIONS:
Device: Soterix Medical mini-CT tDCS stimulator — Patients will have two electrodes applied (one anode, one cathode) administering active (real) or sham (placebo, not real) tDCS stimulation.
  Stimulation will last 20 minutes per day, three days per week, for 5 weeks

SUMMARY:
Transcranial direct current stimulation (tDCS) is a form of non-invasive brain stimulation in which low level electrical currents are applied to the scalp in order to alter brain function. In the present study, tDCS will be administered with the goal of assessing the tolerability and feasibility of this approach to 1) reduce an individual's level of drug craving and 2) provide evidence to support the use of this device by the patient for future unsupervised stimulation in a non-clinical setting.

Research Questions:

* Can tDCS be used successfully to train cocaine addicted individuals for self-administration purposes?
* Can active tDCS be used to decrease drug craving in individuals with cocaine use disorders?
* Does active tDCS outperform sham tDCS in reducing drug craving?

DETAILED DESCRIPTION:
The ultimate goal of this project is to develop a portable neuromodulatory intervention to reduce craving in cocaine addiction. This proposed project is in response to NIH/NIDA's solicitation titled "Development of Portable Neuromodulatory Device for the Treatment of Substance Use Disorders (SUDs)." The present study aims to evaluate the tolerability and feasibility of repeated administration of tDCS to reduce drug craving in individuals with cocaine addiction, with the aim of using these data to support a phase II study and, ultimately, support of approval of usage of this device without clinical supervision.

The specific objectives are:

1. Establish the feasibility and safety of using tDCS to reduce self-reported cravings in individuals addicted to cocaine.
2. Train cocaine addicted individuals to self-administer tDCS (under supervision) to test the feasibility of future home self-administration in this population.

Substance use disorders present a treatment challenge for clinicians, as well as a socioeconomic burden on individuals and society at large. Cocaine use disorder occurs when someone experiences clinically significant impairment caused by the recurrent use of cocaine, including health problems, physical withdrawal with discontinuation of use, persistent/escalating use, and failure to meet major personal, occupational, or educational responsibilities. At present, no FDA approved medicines are available to treat cocaine dependence, and behavioral therapy may be used to treat this addiction, though with limited efficacy. Drug craving (strong obsessions about and/or irresistible urges or compulsions to consume a drug) is a central driving force for perpetuation of substance use and subsequent addiction, as well as relapse after abstinence. Currently, no treatments exist that are targeted at reducing drug craving, which is intrusive and distressing to patients. The prefrontal cortex (PFC) plays an important role inhibiting these intrusive cravings. However, decades of data have shown that PFC activity is impaired in addictions. In this study, our goal is to increase PFC activity with non-invasive neuromodulation. Given the role of the PFC in the processing and regulation of craving behavior, this brain region is a key target for brain stimulation.

This study will recruit individuals with a diagnosis of cocaine use disorder (per DSM-5 criteria) who are receiving treatment for their substance use disorder at Samaritan Daytop Village (SDV) and other similar treatment facilities (e.g., Phoenix House, Mount Sinai's network of hospitals and clinics). Patients will be randomly assigned to receive either active or sham (placebo) tDCS. Participants will receive 20 minutes of stimulation per tDCS day, three days per week for five weeks.

Interviews and neuropsychological testing will be conducted, and self-reported drug craving and addiction severity questionnaires will be used. Follow up cognitive and behavioral assessments will be conducted over a period of 12 months post tDCS stimulation. In addition, participants will be asked to perform EEG, cognitive tasks, and collection of a blood sample to assess genetic/epigenetic patterns.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of cocaine use disorder
* Ability to understand the risks/benefits of the study, provide informed consent and perform tasks as per protocol
* English speaking
* For females of childbearing capacity, current use of a medically acceptable form of birth control

Exclusion Criteria:

* Current or past history of a major neurological disorder (e.g. mental retardation, Parkinson's disease, Lewy body disease, Huntington's disease, MS, ALS, stroke, delirium tremens) or seizures, including those symptoms associated with periods of cocaine withdrawal or abstinence
* History of Axis I disorder, other than substance use disorder, that is associated with psychotic symptoms (e.g. schizophrenia) or neurodevelopmental disorder (e.g., autism)
* Use of medications (current or in the past 6 months) with known CNS effects or which may alter cerebral function, except psychotropics for depression/anxiety/PTSD (e.g. SSRIs)
* Clinically significant unstable medical illness or infection (e.g. HIV, hepatitis, etc.)
* Presence of contraindicated metallic implants or devices which may be impacted by electrical stimulation (e.g. cardiac pacemaker/defibrillator, medication pump, cochlear implant, implanted brain stimulator)
* Head trauma with loss of consciousness for more than 30 minutes
* Pregnancy or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Cocaine Craving from Baseline (Obsessive-Compulsive Cocaine Scale score) | Baseline (pre-tDCS), post-tDCS sessions (approx. week 6), Follow-up (every three months for up to 1 year)
  Craving for cocaine will be assessed with a brief scale composed of 5 items (1, 2, 4, 5, and 13) from the Obsessive-Compulsive Cocaine Scale (OCCS; Vorspan et al., 2012).

SECONDARY OUTCOMES:
Change in Depression symptoms from Baseline (Ham-D score) | Baseline (pre-tDCS), post-tDCS sessions (approx. week 6), Follow-up (every three months for up to 1 year)
  Depression symptoms will be assessed by the Hamilton Rating Scale for Depression (24 item version, HAM-D; Hamilton, 1960).
Change in Anxiety symptoms from Baseline (HAM-A score) | Baseline (pre-tDCS), post-tDCS sessions (approx. week 6), Follow-up (every three months for up to 1 year)
  Anxiety symptoms will be assessed by the Hamilton Rating Scale for Anxiety (HAM-A; Hamilton, 1959).
Change in Quality of Life from Baseline (WHOQOL-BREF score) | Baseline (pre-tDCS), post-tDCS sessions (approx. week 6), Follow-up (every three months for up to 1 year)
  An abbreviated instrument of cross-culturally valid assessment of quality of life of the World Health Organization (WHOQOL-BREF) with 26 questions (WHOQOL Group, 1998; Skevington et al., 2004) yields 4 domains (physical health, psychological, social relationships, and environment) and 2 individually scored items regarding overall perception of quality of life (Q1) and health (Q2). The 4 domain scores are scaled in a way that higher scores stand for higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Datta, PhD, Principal Investigator — Soterix Medical
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batista EK, Klauss J, Fregni F, Nitsche MA, Nakamura-Palacios EM. A Randomized Placebo-Controlled Trial of Targeted Prefrontal Cortex Modulation with Bilateral tDCS in Patients with Crack-Cocaine Dependence. Int J Neuropsychopharmacol. 2015 Jun 10;18(12):pyv066. doi: 10.1093/ijnp/pyv066. PMID 26065432
- [Background] Agarwal S, Pawlak N, Cucca A, Sharma K, Dobbs B, Shaw M, Charvet L, Biagioni M. Remotely-supervised transcranial direct current stimulation paired with cognitive training in Parkinson's disease: An open-label study. J Clin Neurosci. 2018 Nov;57:51-57. doi: 10.1016/j.jocn.2018.08.037. Epub 2018 Sep 5. PMID 30193898
- [Background] Charvet LE, Dobbs B, Shaw MT, Bikson M, Datta A, Krupp LB. Remotely supervised transcranial direct current stimulation for the treatment of fatigue in multiple sclerosis: Results from a randomized, sham-controlled trial. Mult Scler. 2018 Nov;24(13):1760-1769. doi: 10.1177/1352458517732842. Epub 2017 Sep 22. PMID 28937310
- [Background] Charvet L, Shaw M, Dobbs B, Frontario A, Sherman K, Bikson M, Datta A, Krupp L, Zeinapour E, Kasschau M. Remotely Supervised Transcranial Direct Current Stimulation Increases the Benefit of At-Home Cognitive Training in Multiple Sclerosis. Neuromodulation. 2018 Jun;21(4):383-389. doi: 10.1111/ner.12583. Epub 2017 Feb 22. PMID 28225155
- [Background] Moeller SJ, Zilverstand A, Konova AB, Kundu P, Parvaz MA, Preston-Campbell R, Bachi K, Alia-Klein N, Goldstein RZ. Neural Correlates of Drug-Biased Choice in Currently Using and Abstinent Individuals With Cocaine Use Disorder. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 May;3(5):485-494. doi: 10.1016/j.bpsc.2017.11.001. Epub 2017 Nov 11. PMID 29735157
- [Background] Parvaz MA, Moeller SJ, Malaker P, Sinha R, Alia-Klein N, Goldstein RZ. Abstinence reverses EEG-indexed attention bias between drug-related and pleasant stimuli in cocaine-addicted individuals. J Psychiatry Neurosci. 2016 Jul 19;41(5):150358. doi: 10.1503/jpn.150358. Online ahead of print. PMID 27434467
- [Background] Parvaz MA, Moeller SJ, Goldstein RZ. Incubation of Cue-Induced Craving in Adults Addicted to Cocaine Measured by Electroencephalography. JAMA Psychiatry. 2016 Nov 1;73(11):1127-1134. doi: 10.1001/jamapsychiatry.2016.2181. PMID 27603142
- See also: Soterix Medical — https://soterixmedical.com/